CLINICAL TRIAL: NCT03941834
Title: BHV3000-202: Phase 2: A Double-Blind, Placebo Controlled, Crossover Trial of BHV-3000 (Rimegepant) for Treatment Refractory Trigeminal Neuralgia
Brief Title: Trial for Treatment Refractory Trigeminal Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision to discontinue the study based on adjusted clinical development plan. This decision is not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3000-202; C4951014 (Other: Alias Study Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-08 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia, Pain
MeSH Terms: conditions — Trigeminal Neuralgia; Pain | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV3000 (Active Comparator)
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — BHV3000 (rimegepant) 75mg tablet
  Arms: BHV3000
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of BHV3000 compared to placebo for subjects with treatment refractory Trigeminal Neuralgia as measured by a 2-point or greater reduction in the average Numeric Pain Rating Scale between the two-week treatment phases.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a clinical diagnosis of typical or atypical classical trigeminal neuralgia based on the International Classification of Headache Disorders, 3rd edition, beta version.
2. Trigeminal neuralgia symptoms for a minimum of 8 weeks prior to randomization visit.
3. Neuroimaging to exclude another cause for the neuralgia, other than neurovascular compression.

Exclusion Criteria:

1. Subject has a structural lesion on neuroimaging, other than vascular compression of the trigeminal nerve or nerve root that would explain the neuralgia
2. Subject has a clinically evident neurologic deficit on neurologic exam of the cranial nerves
3. Subjects with a history of HIV disease
4. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening
5. Uncontrolled hypertension (high blood pressure) at screening
6. Subject has a current diagnosis of major depression, other pain syndromes, psychiatric conditions (e.g., schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments
7. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has a disease that causes malabsorption
8. Subject has a history or diagnosis of Gilbert's Syndrome or any other active hepatic or biliary disorder
9. The subject has a history or current evidence of any significant and/or unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial
10. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or subjects who have met DSM-V criteria for any significant substance use disorder within the past 12 months from the date of the screening visit
11. Hematologic or solid malignancy diagnosis within 5 years prior to screening. Subjects with a history of localized basal cell or squamous cell skin cancer are eligible for the study if they are cancer-free prior to the screening visit in this study.
12. Hematologic or solid malignancy diagnosis within 5 years prior to screening. Subjects with a history of localized basal cell or squamous cell skin cancer are eligible for the study if they are cancer-free prior to the screening visit in this study.
13. Body mass index >33kg/m²
14. History of gallstones or cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Gilbert Neurology Partners, PLLC/CCT Research, Gilbert, Arizona
  - Center for Neurohealth DBA Kaizen Brain Center, La Jolla, California
  - Imaging Clinic at Stanford Neuroscience Health Center, Palo Alto, California
  - Stanford Hoover Pavilion, Palo Alto, California
  - Stanford Neuroscience Health Center- SNHC Pharmacy, Palo Alto, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Stanford University- CAM Building, Stanford, California
  - SouthCoast Research Center, Miami, Florida
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Johns Hopkins Clinical Outpatient Center, Baltimore, Maryland
  - Johns Hopkins ICTR Clinical Research Unit (CRU), Baltimore, Maryland
  - Clinical Research Professionals, Chesterfield, Missouri
  - Dent Neurosciences Research Center, Amherst, New York
  - Neurological Surgery Practice of Long Island PLCC, Lake Success, New York
  - Neurological Surgery, Lake Success, New York
  - Premier Cardiolog Consultants, Lake Success, New York
  - Premier Cardiolog Consultants, New Hyde Park, New York
  - Premier Cardiology Consultants, New Hyde Park, New York
  - North Suffolk Neurology, PC, Port Jefferson Station, New York
  - Neurology Diagnostics Inc., Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 phases in the study: double blind treatment (DBT) phase followed by open label extension (OLE) phase. Participants after completing DBT phase could enter OLE phase if the Principal Investigator (PI) believed open-label treatment offered an acceptable risk-benefit profile. A total of 65 participants with refractory trigeminal neuralgia (TN) were enrolled in the study.
Pre-assignment Details: Out of 65 participants, only 30 were randomized in DBT phase, and 35 participants were not randomized (screen failure [28], sponsor decision [1], medical monitor decision [1], physician decision [1], withdrawal of consent [4]).
Groups:
- DBT Phase: Placebo Then Rimegepant (BHV-3000): Participants included in this arm were randomized to first sequence. Participants in first treatment period received placebo (matched to rimegepant) orally once daily (QD) for 2 weeks and in second treatment period received rimegepant 75 milligram (mg) immediate release (IR) tablet orally QD for 2 weeks. Treatment periods were separated by a washout period of 7 days.
- DBT Phase: Rimegepant Then Placebo: Participants in first treatment period received rimegepant 75 mg IR tablet orally QD for 2 weeks and in second period received placebo (matched to rimegepant) QD for 2 weeks. Treatment periods were separated by a washout period of 7 days.
- OLE Phase: Rimegepant: Participants who completed DBT phase, were eligible per PI judgment and agreed to enter OLE phase, received rimegepant 75 mg Orally disintegrating tablet (ODT) QD for 12 weeks in OLE phase.
Period: DBT Phase: 1st Treatment Period (2Weeks)
Arm/Group | DBT Phase: Placebo Then Rimegepant (BHV-3000) | DBT Phase: Rimegepant Then Placebo | OLE Phase: Rimegepant
Started | 15 | 15 | 0
Treated | 15 | 14 | 0
Completed | 14 | 14 | 0
Not Completed | 1 | 1 | 0
Not completed — Randomized but not treated | 0 | 1 | 0
Not completed — Non compliance | 1 | 0 | 0
Period: DBT Phase: Washout Period (7 Days)
Arm/Group | DBT Phase: Placebo Then Rimegepant (BHV-3000) | DBT Phase: Rimegepant Then Placebo | OLE Phase: Rimegepant
Started | 14 | 14 | 0
Completed | 14 | 14 | 0
Not Completed | 0 | 0 | 0
Period: 2nd Treatment Period (2Weeks)
Arm/Group | DBT Phase: Placebo Then Rimegepant (BHV-3000) | DBT Phase: Rimegepant Then Placebo | OLE Phase: Rimegepant
Started | 14 | 14 | 0
Completed | 14 | 14 | 0
Not Completed | 0 | 0 | 0
Period: OLE Phase (12 Weeks)
Arm/Group | DBT Phase: Placebo Then Rimegepant (BHV-3000) | DBT Phase: Rimegepant Then Placebo | OLE Phase: Rimegepant
Started | 0 (This arm is for DBT phase. Participants only for OLE Phase recorded in this period.) | 0 (This arm is for DBT phase. Participants only for OLE Phase recorded in this period.) | 13 (Eligible participants entered OLE phase after completing DBT phase.)
Completed | 0 | 0 | 9
Not Completed | 0 | 0 | 4
Not completed — Study terminated by sponsor | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Sponsor decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of double-blind study drug in DBT phase and OLE phase. Participants in DBT and OLE phases are not exclusive. Eligible participants from DBT phase entered OLE phase after completing treatment in DBT phase.
Groups:
- DBT: Placebo Then Rimegepant: Participants in first treatment period received placebo (matched to rimegepant) QD for 2 weeks and in second treatment period received rimegepant 75 mg IR tablet orally QD for 2 weeks.
- DBT Phase: Rimegepant Then Placebo: Participants in first treatment period received rimegepant 75 mg IR tablet orally QD for 2 weeks and in second treatment period received placebo (matched to rimegepant) QD for 2 weeks.
- OLE Phase: Rimegepant: Participants received rimegepant 75 mg ODT QD for 12 weeks in OLE phase.
- Total: Total of all reporting groups
Arm/Group | DBT: Placebo Then Rimegepant | DBT Phase: Rimegepant Then Placebo | OLE Phase: Rimegepant | Total
Number analyzed (Participants) | 15 | 14 | 13 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Number Analyzed for DBT Phase and OLE Phase = number of participants analyzed for reporting arms for respective phases. Participants in DBT and OLE phases are not exclusive.
  Years
    DBT Phase: number analyzed (Participants) | 15 | 14 | 0 | 29
    DBT Phase | 57.9 (13.05) | 66.2 (14.61) |  | 61.9 (14.21)
    OLE Phase: number analyzed (Participants) | 0 | 0 | 13 | 13
    OLE Phase |  |  | 61.8 (17.83) | 61.8 (17.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number Analyzed for DBT Phase and OLE Phase = number of participants analyzed for reporting arms for respective phases. Participants in DBT and OLE phases are not exclusive.
  Participants
    DBT Phase: number analyzed (Participants) | 15 | 14 | 0 | 29
    DBT Phase: Female | 11 | 10 |  | 21
    DBT Phase: Male | 4 | 4 |  | 8
    OLE Phase: number analyzed (Participants) | 0 | 0 | 13 | 13
    OLE Phase: Female |  |  | 10 | 10
    OLE Phase: Male |  |  | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed for DBT Phase and OLE Phase= number of participants analyzed for reporting arms for respective phases. Participants in DBT and OLE phases are not exclusive.
  Participants
    DBT Phase: number analyzed (Participants) | 15 | 14 | 0 | 29
    DBT Phase: Hispanic or Latino | 3 | 4 |  | 7
    DBT Phase: Not Hispanic or Latino | 12 | 10 |  | 22
    DBT Phase: Unknown or Not Reported | 0 | 0 |  | 0
    OLE Phase: number analyzed (Participants) | 0 | 0 | 13 | 13
    OLE Phase: Hispanic or Latino |  |  | 5 | 5
    OLE Phase: Not Hispanic or Latino |  |  | 8 | 8
    OLE Phase: Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number Analyzed for DBT Phase and OLE Phase = number of participants analyzed for reporting arms for respective phases. Participants in DBT and OLE phases are not exclusive.
  Participants
    DBT Phase: number analyzed (Participants) | 15 | 14 | 0 | 29
    DBT Phase: American Indian or Alaska Native | 0 | 0 |  | 0
    DBT Phase: Asian | 0 | 0 |  | 0
    DBT Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    DBT Phase: Black or African American | 3 | 1 |  | 4
    DBT Phase: White | 12 | 12 |  | 24
    DBT Phase: More than one race | 0 | 0 |  | 0
    DBT Phase: Unknown or Not Reported | 0 | 1 |  | 1
    OLE Phase: number analyzed (Participants) | 0 | 0 | 13 | 13
    OLE Phase: American Indian or Alaska Native |  |  | 0 | 0
    OLE Phase: Asian |  |  | 0 | 0
    OLE Phase: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
    OLE Phase: Black or African American |  |  | 2 | 2
    OLE Phase: White |  |  | 10 | 10
    OLE Phase: More than one race |  |  | 0 | 0
    OLE Phase: Unknown or Not Reported |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Daily Pain Score on Numeric Pain Rating Scale (NPRS) at 2 Week Treatment Phase: DBT Phase
Description: NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable), higher scores represent worse pain. Participants daily recorded their average pain level over a 24-hour period on NPRS. Pain score was the average of the daily 11-point NPRS recorded within each period. Average of pain score on NPRS according to treatment received in first or second treatment period of DBT phase are used for evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline (before dose on Day 1), 2 Weeks Treatment
Population: Modified intent-to-treat (mITT) analysis set included randomized participants who received at least 1 dose of study therapy and provided a baseline and at least one post-baseline efficacy assessment in each sequence. Here, "Number of Participants Analyzed" signifies number of participants in mITT set, per treatment (pooled) received either in first or second treatment period of DBT phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- DBT Phase: Pooled Rimegepant: Participants who received rimegepant 75 mg IR tablet in treatment period 1 or 2 of DBT phase.
- DBT Phase: Pooled Placebo: Participants who received placebo matched to rimegepant in treatment period 1 or 2 of DBT phase.
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale | -.5 [-1.1 to -.1] | -1.2 [-1.8 to -0.6]
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis were performed using a mixed model with fixed effects for treatment, period and sequence; baseline NPRS as a covariate; and participant as a random effect; Test type: Other; Least square (LS) mean difference = 0.7, 95% CI 2-sided [0.1 to 1.2]

2. Secondary Outcome: Number of Participants With All-Causality Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Study Drug Discontinuation and Treatment Related AEs: DBT Phase
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect other important medical events. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness to drug was assessed by investigator.
Time Frame: DBT Phase: Day 1 of dosing up to last day of dosing (up to 5 weeks)
Population: DBT treated set consisted of participants in the treated analysis set who took >= 1 dose of DB study drug (rimegepant or placebo), i.e., non-missing study drug start date. Here, "Number of Participants Analyzed" signifies number of participants in DBT treated set, per treatment (pooled) received either in first or second treatment period of DBT phase.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 29
Participants
  SAEs | 0 | 0
  AEs Leading to Study Drug Discontinuation | 0 | 0
  Treatment Related AEs | 4 | 0

3. Secondary Outcome: Number of Participants With Any Change From Baseline in Sheehan Suicidality Tracking Scale (S-STS) Scores: DBT Phase
Description: S-STS is a scale that assesses the seriousness of suicidality phenomena on a 5-point Likert-type scale (0 to 4) ranging from "not at all" (0) to "extremely" (4), where higher scores signify suicidal tendency. In this outcome measure, number of participants who had any change in S-STS score from baseline to end of treatment are reported according to the treatment received in first or second treatment period of DBT phase.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 29
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities: DBT Phase
Description: ECG abnormalities included were a Corrected QT interval exceeding 470 milliseconds (QTc calculated using the Frederica method), left bundle branch block, right bundle branch block with a QRS duration of 150 milliseconds or more, and intraventricular conduction defect with a QRS duration equal to or greater than 150 milliseconds. Clinical significance in ECG abnormalities was judged by investigator.
Time Frame: DBT Phase: Day 1 of dosing up to last day of dosing (up to 5 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 29
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: DBT Phase
Description: Laboratory abnormalities included 1)Hematology: hemoglobin, hematocrit, platelets, complete blood count with differential and absolute neutrophil count; 2)Serum chemistry: sodium, potassium, chloride, calcium, alanine aminotransferase, aspartate aminotransferase, lactate dehydrogenase, alkaline phosphatase, gamma-glutamyl transferase, phosphorus, bicarbonate, creatine phosphokinase, total protein, albumin, total bilirubin, glucose, creatinine, blood urea nitrogen, uric acid, total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides, folate, hemoglobin A1C, pancreatic amylase or lipase, thyroid-stimulating Hormone, thyroxine; 3)Urinalysis: macroscopic examination, pH, specific gravity, ketones, nitrites, urobilinogen, leukocyte esterase, protein, glucose, occult blood; 4)Liver function tests: alanine aminotransferase, aspartate aminotransferase, total bilirubin, alkaline phosphatase. Clinical significance in laboratory abnormalities was judged by investigator.
Time Frame: DBT Phase: Day 1 of dosing up to last day of dosing (up to 5 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 29
Participants | 0 | 0

6. Secondary Outcome: Change From Baseline in Penn Facial Pain Scale-Revised (Penn-FPS-R) Total Score at 2 Week Treatment Phase: DBT Phase
Description: Penn-FPS-R: a 12-item scale, utilized to evaluate the impact of TN pain on health-related quality of life and daily activities. Each 12 items ranged from 0 (does not interfere) to 10 (completely interferes). Penn-FPS-R total score was calculated by adding scores of all items and had a score range of (does not interfere) 0 to 120 (completely interferes).Higher Penn-FPS-R total scores signifies worse condition. Participants were asked to complete the Penn-FPS-R at the beginning and end of each treatment period. Average of total Penn-FPS-score according to treatment received in first or second treatment period of DBT phase are used in evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: mITT analysis set included randomized participants who received at least 1 dose of study therapy and provided a baseline and at least one post-baseline efficacy assessment in each sequence. Here, "Number of Participants Analyzed" signifies number of participants in mITT set, per treatment (pooled) received either in first or second treatment period of DBT phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale | -14.2 [-22.2 to -6.2] | -16.6 [-24.6 to -8.6]
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis was performed using a mixed model with fixed effects for treatment, period and sequence; baseline Penn-FPS-R as a covariate; and participant as a random effect; Test type: Other; LS mean difference = 2.4, 95% CI 2-sided [-6.8 to 11.5]

7. Secondary Outcome: Change From Baseline in Pain Disability Index Total Score at 2 Week Treatment Phase: DBT Phase
Description: Pain disability index measures the extent of disruption in a participant's daily life caused by pain, utilizing a 7-item scale scored on an 11-point Likert Scale, where "0" denotes "no disability," and "10" indicates "worst disability". Higher scores signify worse outcome. Pain disability index total score was calculated by adding scores of all the 7 items and had a score range of 0 to 70. Higher pain disability index total scores signifies worse condition. Participants were instructed to complete the pain disability index at the beginning and end of each treatment period. Average of pain disability index total scores according to treatment received in first or second treatment period of DBT phase are used for evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale | -7.8 [-12.6 to -2.9] | -9.3 [-14.2 to -4.5]
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis was performed using a mixed model with fixed effects for treatment, period and sequence; baseline pain disability index as a covariate; and participant as a random effect; Test type: Other; LS Mean Difference = 1.5, 95% CI 2-sided [-3.8 to 6.9]

8. Secondary Outcome: Patient Global Impression of Change Scale (PGI-C) Score at 2 Week Treatment Phase: DBT Phase
Description: PGI-C is a participant-reported scale utilized to evaluate the improvement or deterioration of the participant's current illness status compared to the baseline visit. Participants were asked to rate a change in their overall disease condition on a 7-point scale, ranging from 1 (no change) to 7 (a great deal better). Higher PGI-C scores signify better outcome. PGI-C assessments were conducted at the beginning and end of each treatment phase. Average of PGI-C score according to treatment received in first or second treatment period of DBT phase are used in evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale | 3.0 [2.3 to 3.8] | 3.1 [2.4 to 3.8]
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis was performed using a mixed model with fixed effects for treatment, period and sequence; and participant as a random effect; Test type: Other; LS Mean Difference = -0.1, 95% CI 2-sided [-0.7 to 0.5]

9. Secondary Outcome: Change From Baseline in Average Worst Pain Score on NPRS at 2 Week Treatment Phase: DBT Phase
Description: NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable), higher scores represent worse pain. Participants daily recorded their worst pain rating over a 24-hour period on NPRS. Average of worst pain NPRS score according to treatment received in first or second treatment period of DBT phase are used in evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale | -0.6 [-1.3 to 0.1] | -1.3 [-2.0 to -0.6]
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis was performed using a mixed model with fixed effects for treatment, period and sequence; baseline NPRS as a covariate; and participant as a random effect; Test type: Other; LS Mean Difference = 0.7, 95% CI 2-sided [0.1 to 1.4]

10. Secondary Outcome: Percentage of Participants With >= 2 Point Reduction From Baseline in Average Daily Pain Score on NPRS at 2 Week Treatment Phase: DBT Phase
Description: NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable), higher scores represent worse pain. Participants daily recorded their average pain level over a 24-hour period. Pain score was the average of the daily 11-point NPRS recorded within each period. Average of pain score on NPRS according to treatment received in first or second treatment period of DBT Phase are used in evaluation of the outcome measure.
Time Frame: DBT Phase: Baseline, 2 Weeks Treatment
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo
Number analyzed (Participants) | 28 | 28
Percentage of participants | 10.7 | 35.7
Statistical Analysis 1: Comparison: DBT Phase: Pooled Rimegepant vs DBT Phase: Pooled Placebo; Analysis was performed using a logistic regression model, including fixed effects for treatment, sequence, period and baseline NPRS score as a covariate; Test type: Other; Odds Ratio (OR) = 12.6, 95% CI 2-sided [0.7 to 229.6]

ADVERSE EVENTS:
Time Frame: Day 1 up to 2 weeks of follow up post-last dose in the study (Maximum up to 19 weeks)
Description: Treated analysis set evaluated.
Groups:
- DBT Phase/ Treatment Sequence 1/ Period 1: Placebo: Participants included in this arm were randomized to first sequence to receive placebo (matched to rimegepant) orally QD for 2 weeks in Period 1.
- DBT Phase/ Treatment Sequence 1/ Period 2: Rimegepant: Participants included in this arm were randomized to first sequence to receive rimegepant 75 mg IR tablet orally QD for 2 weeks in Period 2.
- DBT Phase/ Treatment Sequence 2/ Period 1: Rimegepant: Participants included in this arm were randomized to second sequence to receive rimegepant 75 mg IR tablet orally QD for 2 weeks in Period 1.
- DBT Phase/ Treatment Sequence 2/ Period 2: Placebo: Participants included in this arm were randomized to second sequence to receive placebo (matched to rimegepant) orally QD for 2 weeks in Period 2.
Arm/Group | DBT Phase/ Treatment Sequence 1/ Period 1: Placebo | DBT Phase/ Treatment Sequence 1/ Period 2: Rimegepant | DBT Phase/ Treatment Sequence 2/ Period 1: Rimegepant | DBT Phase/ Treatment Sequence 2/ Period 2: Placebo | DBT Phase: Pooled Rimegepant | DBT Phase: Pooled Placebo | OLE Phase: Rimegepant
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/14 | 0/28 | 0/29 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14 | 0/14 | 0/28 | 0/29 | 0/13
Other Adverse Events (participants affected / at risk) | 1/15 | 3/14 | 3/14 | 0/14 | 6/28 | 1/29 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBT Phase/ Treatment Sequence 1/ Period 1: Placebo (N=15) | DBT Phase/ Treatment Sequence 1/ Period 2: Rimegepant (N=14) | DBT Phase/ Treatment Sequence 2/ Period 1: Rimegepant (N=14) | DBT Phase/ Treatment Sequence 2/ Period 2: Placebo (N=14) | DBT Phase: Pooled Rimegepant (N=28) | DBT Phase: Pooled Placebo (N=29) | OLE Phase: Rimegepant (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 2 | 0 | 3 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03941834/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03941834/SAP_001.pdf